CLINICAL TRIAL: NCT04386369
Title: Evaluation of Airway Pressure Release Ventilation on Oxygenation in Acute Respiratory Distress Syndrome in Adult Patients With COVID-19 Pneumonia
Brief Title: Evaluation of Airway Pressure Release Ventilation in COVID-19 ARDS
Acronym: APRV-COVID19
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI076
Record Dates: First submitted 2020-04-14; First posted 2020-05-13 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-04

CONDITIONS: ARDS; COVID19
Keywords: Airway Pressure Release Ventilation; Intensive Care Unit; SARS-CoV-2; APRV; Acute respiratory failure
MeSH Terms: conditions — COVID-19 | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Airway Pressure Release Ventilation: Patients with COVID-19 ARDS requiring invasive mechanical ventilation in ICU, on Volume Assist Control ventilation (VAC) or Pressure Assist Control (PAC), are switched to airway pressure ventilation (APRV). If APRV doesn't lead to improvement in oxygenation the ventilatory mode is switched back to VAC or PAC ventilatory mode.
  Interventions: Other: Airway pressure release ventilation

INTERVENTIONS:
Other: Airway pressure release ventilation — Ventilator management strategy

SUMMARY:
The 2020 pandemic of the coronavirus (SARS-CoV2) has lead to an increase in ARDS cases requiring invasive mechanical ventilation in the ICU (Intensive Care Unit).

The investigators hypothesize that airway pressure release ventilation (APRV) could be beneficial in patients with ARDS secondary to SARS-COV2 viral pneumonia.

DETAILED DESCRIPTION:
Lung protective mechanical ventilation is the cornerstone of ARDS management, reducing the work of respiratory muscles and optimizing gas exchange. However, it can be the source of deleterious effects, grouped under the terms of ventilator induced lung injury (VILI) and ventilator induced diaphragm dysfunction.

The protective ventilatory strategy has led to a significant improvement in the prognosis of ARDS patients, by reducing the volume of the air and oxygen mixture (lower tidal volume) delivered to the lungs and thus reducing the pulmonary stress and strain. However, this protective ventilation usually requires deep sedation and neuromuscular blockade to avoid deleterious patient-ventilator asynchrony.

Airway Pressure Release Ventilation (APRV) has been proposed to reduce patient-ventilator asynchrony and reduce the VILI. The operating principles of APRV are based on the presence of two pressure levels that are kept constant. Spontaneous breathing is possible at any time at both pressure levels if the patient is not deeply sedated or under neuromuscular blockade.

The investigators hypothesize that APRV mode could be beneficial on oxygenation and respiratory work in patients with ARDS secondary to SARS-COV2 viral pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated in Nancy University Hospital between 01/04/2020 and 31/06/2020 for COVID-19 ARDS, requiring invasive ventilation
* Trial of airway pressure release ventilation during the ICU stay

Exclusion Criteria:

* Patients requiring veno-venous ECMO
* Patients unable to complete the 6-hour APRV trial due to poor tolerance : SpO2 decrease < 90% on FiO2 70%, haemodynamic instability (MAP < 65mmhg without vasopressors, or 0.5 mg/h increase in norepinephrine, ventilator asynchrony (respiratory rate >35), hypercapnia (pH < 7,25 or PaCO2 >60mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to the Intensive Care Unit for treatment of COVID-19 related acute respiratory failure.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients improving PaO2/FiO2 ratio at 6 hours of APRV | 6 hours after starting APRV
  Increase of at least 20% of the PaO2/FiO2 ratio

SECONDARY OUTCOMES:
Number of interventions on ventilator settings | 6 hours after starting APRV
  Number of interventions by the physician on APRV settings
Change in mean blood pressure | 6 hours after starting APRV
  Variations of blood pressure in millimeters of mercury
Change in heart rate | 6 hours after starting APRV
  Variations of heart rate in beats per minute
Changes in catecholamine doses | 6 hours after starting APRV
  Variations of catecholamine doses in milligrams per hours
Changes in static compliance at the end of 6 hours of APRV | 6 hours after starting APRV
  Static compliance (Cstat) defined as : Cstat = (VT/(Pplat-PEPtot)) Tidal Volume (VT), Plateau pressure (Pplat) and Total Positive End-expiratory Pressure (PEEPtot)
Variations of minute ventilation | 6 hours after starting APRV
  Minute ventilation in liters per minute
Changes in static compliance 4 hours after stopping APRV | 4 hours after starting APRV
  Static compliance (Cstat) defined as : Cstat = (VT/(Pplat-PEPtot)) Tidal Volume (VT), Plateau pressure (Pplat) and Total Positive End-expiratory Pressure (PEEPtot)
Proportion of patients with a decrease of the PaO2/FiO2 ratio | 4 hours after stopping APRV
  Percentage of patients with a decrease of the PaO2/FiO2 ratio

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu Koszutski, MD, Principal Investigator — CHRU de NANCY, Médecine Intensive et Réanimation Brabois
Locations (1):
- Centre Hospitalier Régional Universitaire de Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou Y, Jin X, Lv Y, Wang P, Yang Y, Liang G, Wang B, Kang Y. Early application of airway pressure release ventilation may reduce the duration of mechanical ventilation in acute respiratory distress syndrome. Intensive Care Med. 2017 Nov;43(11):1648-1659. doi: 10.1007/s00134-017-4912-z. Epub 2017 Sep 22. PMID 28936695
- [Background] Nieman GF, Al-Khalisy H, Kollisch-Singule M, Satalin J, Blair S, Trikha G, Andrews P, Madden M, Gatto LA, Habashi NM. A Physiologically Informed Strategy to Effectively Open, Stabilize, and Protect the Acutely Injured Lung. Front Physiol. 2020 Mar 19;11:227. doi: 10.3389/fphys.2020.00227. eCollection 2020. PMID 32265734